CLINICAL TRIAL: NCT06003933
Title: Inter-semispinal Plane (ISP) Block for Postoperative Analgesia Following Cervical Spine Surgery: A Prospective Randomized Controlled Trial
Brief Title: Inter-semispinal Plane Block and Cervical Spine Surgery
Acronym: ISPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser S Mostafa, MD (Other)
Responsible Party: Sponsor-Investigator, Yasser S Mostafa, MD, Lecturer of anesthesia, Fayoum University Hospital
Organization: Fayoum University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: m644
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Post Operative Pain; Cervical Spine Instability
Keywords: inter-semispinal plane block; Cervical spine surgery; Postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Lidocaine; Ultrasonography; Needles

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated into either of the two groups using computer generated sequence and concealed in sealed opaque envelopes.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): patients received general anesthesia only.
- ISP group (Experimental): patients received bilateral ultrasound guided inter-semispinal plane (ISP) block at the level of C5 using 10 ml of 0.25% bupivacaine and 10ml xylocaine on each side to reduce the toxicity
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Lidocaine Hydrochloride; Device: Ultrasound; Device: Needle

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — 10 ml of 0.25% bupivacaine on each side of cervical region at C5
  Other Names: 0.25% bupivacaine HCL
  Arms: ISP group
Drug: Lidocaine Hydrochloride — 10ml xylocaine on each side of cervical region at C5
  Other Names: Xylocaine
  Arms: ISP group
Device: Ultrasound — The same anesthesiologist who is experienced in US guided regional anesthesia will perform the block.The five-layered posterior cervical muscles were identified at the level of C5 with a 6-15-MHz linear probe oriented in the transverse plane (SonoSite Edge, Bothell, Washington). The fifth cervical spine was counted from the C7 spinous process with the probe sliding cranially.
  Arms: ISP group
Device: Needle — the needle (22- G, 50-mm block needle (Visioplex, Vygon) was introduced in-plane through the skin and advanced into the fascial plane between the semispinalis cervicis and semispinalis capitis muscles. After negative aspiration for blood, 20 ml of bupivacaine 0.25% was injected5.
  Arms: ISP group

SUMMARY:
The inter-semispinal plane (ISP) block is a novel ultrasound-guided technique that involves local anesthetic injection into the fascial plane between the semispinalis cervicis and semispinalis capitis muscles with subsequent block of the dorsal rami of the cervical spinal nerves and hence can get adequate postoperative analgesia.

The authors hypothesized that ISP block can reduce the postoperative analgesic consumption in patients undergoing posterior cervical spine surgeries.

The aim of this study is to evaluate the analgesic efficacy of ISP block in patients undergoing posterior cervical spine surgery.

DETAILED DESCRIPTION:
This study will be performed in the in the Fayoum University hospital after the local Institutional Ethics Committee and local institutional review board approval. The study design will be double-blind randomized controlled study . A detailed informed consent will be signed by the eligible patients before recruitment and randomization.

Patients were randomly allocated into two groups using computer generated sequence and concealed in sealed opaque envelopes.

Control group (C): patients received general anesthesia only. Inter-semispinal plane (ISP) block group: patients received bilateral ultrasound guided ISP block at the level of C5.

All patients will be assessed Preoperative VAS score then premedicated orally with midazolam 0.5 mg/kg 30 min prior to surgery. All patients were monitored by 5 lead ECG, pulse oximetry, non-invasive blood pressure and capnography and an intravenous (IV) access will be established.

The technique of general anesthesia will be standardized for all patients. General anesthesia will be induced by intravenous (IV) 2 mg/kg propofol and 1 μg/kg fentanyl induction. After IV atracurium 0.5 mg/kg, orotracheal intubation was performed. Anesthesia will be maintained with isoflurane (1.2%-1.5%) in oxygen-air mixture (50%-50%). Muscle relaxation will be maintained during the procedure with atracurium in increments.

After induction of general anesthesia, ISP blocks will be performed in the allocated group with the patient in the prone position. In both groups, the treating anesthesiologist left the operating room while another anesthesiologist experienced in ultrasound guided nerve block techniques; with no subsequent role in the study; either performed the ISP blocks in the ISP group, or just prepared the skin and scanned the site of the block using the ultrasound probe in the control group. Fifteen minutes will be awaited in all patients before the surgical procedure was allowed to start.

fentanyl 0.5 μg/kg IV will be administered in case of inadequate analgesia as indicated by >20% increase in heart rate or mean arterial blood pressure. Total intraoperative fentanyl consumption will be recorded.

All anesthetics will be discontinued at the end of the surgical procedure. Extubation will be performed when spontaneous breathing was adequate and following prompt reversal using 0.05 mg/kg of neostigmine and 0.02 mg/kg of atropine. At the end of surgery, paracetamol 1 g will be administered IV to be repeated every 6 h postoperatively. Patients will be transferred to the PACU where HR, respiratory rate, SpO2 and systolic, diastolic and mean arterial blood pressure were monitored.

Sample size was calculated using G* Power 3.1.7.9 software program. Calculation of the sample size was based on the VAS value measured at different time points. Based on the results of a study by Mostafa et al, the authors calculated the sample size to be able to detect a difference in VAS score of 10 points with an effect size of 0.8. Using the previous data, at least 23 patients in each group were required to detect a significance difference in the postoperative pethidine consumption at α value of 0.05 and study power of 90%. The authors decided to recruit 25 patients in each group to compensate for any possible withdrawals. The sample size calculation was based on a 2-sample independent t-test (2-sided)

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II undergoing elective posterior cervical spine surgery

Exclusion Criteria:

* Patient refusal
* Patients with any contraindication to regional anesthesia (e.g. local infection, coagulation abnormality)
* Known allergy to local anesthetics
* Previous cervical disc surgery or fixation
* Mental disorders
* Drug or alcohol abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
postoperative rescue pethidine consumption | 48 hours after operation
  in milligram

SECONDARY OUTCOMES:
Postoperative visual analog pain score (VAS score) | 4 hours postoperatively
  0 to 10 scale as 0: no pain and 10:worst degree of pain
Postoperative visual analog pain score (VAS score) | 8 hours postoperatively
  0 to 10 scale as 0: no pain and 10:worst degree of pain
Postoperative visual analog pain score (VAS score) | 12 hours postoperatively
  0 to 10 scale as 0: no pain and 10:worst degree of pain
Postoperative visual analog pain score (VAS score) | 24 hours postoperatively
  0 to 10 scale as 0: no pain and 10:worst degree of pain
Postoperative visual analog pain score (VAS score) | 48 hours postoperatively
  0 to 10 scale as 0: no pain and 10:worst degree of pain
time to first rescue analgesic request | 1 minute after requiring analgesics
  in milligram
Intraoperative fentanyl consumption | 1 minute after surgery.
  in microgram
Occurrence of postoperative nausea | 2 hours after operation
  yes or no
Occurrence of postoperative vomiting | 2 hours after operation
  yes or no
Occurrence of postoperative pruritis | 2 hours after operation
  yes or no

OTHER OUTCOMES:
Age | 1 hour preoperatively
  in years
body mass index | 1 hour preoperatively
  kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Shawky, MD, Study Director — Fayoum University
Locations (1):
- Fayoum University Hospital, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurd MF, Kreitz T, Schroeder G, Vaccaro AR. The Role of Multimodal Analgesia in Spine Surgery. J Am Acad Orthop Surg. 2017 Apr;25(4):260-268. doi: 10.5435/JAAOS-D-16-00049. PMID 28291143
- [Background] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Ay AN, Celik EC, Karaavci NC. Postoperative Analgesic Efficacy of the Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Lumbar Spinal Decompression Surgery: A Randomized Controlled Study. World Neurosurg. 2019 Jun;126:e779-e785. doi: 10.1016/j.wneu.2019.02.149. Epub 2019 Mar 8. PMID 30853517
- [Background] Lumawig JM, Yamazaki A, Watanabe K. Dose-dependent inhibition of diclofenac sodium on posterior lumbar interbody fusion rates. Spine J. 2009 May;9(5):343-9. doi: 10.1016/j.spinee.2008.06.455. Epub 2008 Sep 14. PMID 18790686